CLINICAL TRIAL: NCT02419885
Title: Evaluation of Result and Influence Factors on Composite Graft in Fingertip Amputation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUH-IRB
Record Dates: First submitted 2015-04-06; First posted 2015-04-17 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 1990-12

CONDITIONS: Pinprick Sensation Diminished; Amputation, Traumatic; Pain
Keywords: finger amputation; composite graft; adipo-fascia flap
MeSH Terms: conditions — Somatosensory Disorders; Amputation, Traumatic; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Fingertips facilitate smooth motor activity, precise sensation, and the delicate movement of the hands and have an aesthetic function. Fingertip injuries are defined as injuries occurring distal to the insertion of the flexor and extensor tendons. These injuries are one of the most common trauma injuries presented in acute care settings, accounting for approximately 4.8 million emergency department visits per year in the United States.(1) Fingertip amputations may not constitute the majority among these fingertip injuries but can have a complex spectrum of injury. In these cases, the reconstruction methodologies focus on preserving the digital length, ensuring adequate soft tissue coverage, preserving the nail structure, achieving a well-contoured and painless fingertip, and restoring durable and sensate skin.

There are so many factor that influence the result of composite graft in distal finger tip amputation. Investigators will collected the data including the size of amputee , shape, level of amputation, mechanism of amputation, if hyperbaric oxygen therapy, operation procedures.

DETAILED DESCRIPTION:
Fingertip amputations underwent

1. modified composite grafting with pulp Adipo-fascia advance flap
2. composite graft
3. revision amputation was collected in this study

Follow-up was arranged in out-patient department, including:

type of amputation ( Hirase classification, ) 2-point discrimination test, DASH(Disabilities of the Arm, Shoulder, and Hand) outcome measure, graft survival, pain evaluation with visual Analog scale other associated treatment such as hyperbaric oxygen therapy length of finger shortening at 6 month after operation

ELIGIBILITY:
Inclusion Criteria:

* February 1990 and June 2015, patients received composite graft in fingertip amputation

Exclusion Criteria:

* patients refused to participate the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective chart review study. Patients were collected since 1990,
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
graft survival | postoperatively after 6 weeks
  composite graft survival rate

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | postoperatively 24 weeks
  hand function evaluation
subjective self-evaluation questionnaire | postoperatively 24 weeks
  subjective self-evaluation of finger looking
length of finger shortening | postoperatively 24 weeks
  finger length

CONTACTS AND LOCATIONS:
Overall Officials: huang shu-hung, MD, Study Chair — Division of Plastic Surgery, Department of Surgery, Kaohsiung Medical University Hospital
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan, Taiwan